CLINICAL TRIAL: NCT06231758
Title: The AMPK Modulator Metformin as a Novel Adjunct to Conventional Therapy in Patients With Knee Osteoarthritis
Brief Title: Metformin Safety and Efficacy in Osteoarthritis.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Teaching assisstant, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Menofya 1247
Record Dates: First submitted 2024-01-20; First posted 2024-01-30 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Osteo Arthritis Knee
MeSH Terms: interventions — Celecoxib; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): 35 patients will receive celecoxib 200 mg capsule plus placebo tablets
  Interventions: Drug: Celecoxib 200mg
- Comparative group (Active Comparator): 35 patients will receive celecoxib 200 mg capsule plus 1000 mg metformin daily
  Interventions: Drug: Celecoxib 200mg; Drug: Metformin

INTERVENTIONS:
Drug: Celecoxib 200mg — Celecoxib is a nonsteroidal anti-inflammatory drug (NSAID) used to treat mild to moderate pain and help relieve symptoms of arthritis (eg, osteoarthritis, rheumatoid arthritis, or juvenile rheumatoid arthritis), such as inflammation, swelling, stiffness, and joint pain.
Drug: Metformin — Metformin (MET), a traditional antdiabetic drug, exerts glucose-lowering effect by activating AMPK since it is a critical enzyme in lipid and glucose metabolism
  Arms: Comparative group

SUMMARY:
Knee osteoarthritis (OA) is a chronic, painful disease associated with considerable morbidity, costs and disability. It is estimated that over a third of people aged over 60 have radiographic knee OA2 and over 50% of these with knee OA will go on to have a total knee replacement in their lifetime. At present there are no licensed treatments that alter disease progress and management is primarily concerned with symptom control to retain or improve joint function, although a trial of strontium ranelate showed promising results.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis Patients recruited were between 30 to 60 years of age.
* X-ray confirmed Kellgren-Lawrence grade II or III severity primary tibiofemoral OA according to the American College of Rheumatology criteria.

Exclusion Criteria:

Patients with age less than 30 years or more than 60 years Patients Presented with active concomitant gastroduodenal disorders, hepatic and renal impairment within last 30 days prior to receiving the study drug Patients Were diagnosed to have any inflammatory arthritis, gout or acute trauma of the knee, hip or spine; accompanying OA of the hip of sufficient severity to interfere with the functional assessment of the knee Patients had previous or ongoing treatment with oral SYSDOA (e.g., glucosamine sulphate, chondroitin sulphate, diacerein, piascledine), anti-depressants, tranquillisers, antacids or antibiotics; were having active cardiac lesion or hypertension, were pregnant females and those who were planning their pregnancy during the study Patients having a known hypersensitivity to the used medications Patients have persistent diarrhoea or laxative use; severe gastrointestinal disorders, severe obesity, severe parenchymal organ disease, or anaemia (haemoglobin< 10.0 g/ dl or haematocrit < 30%).

Patients who received oral, intramuscular, intraarticular or soft tissue injections of corticosteroids within last eight weeks before receiving the first dose of the study medication or had undergone joint lavage and arthroscopic procedures in the previous 6 months, were also excluded.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy end point will be the change of Visual Analogue Scale (VAS) pain score from baseline to post treatment. | 3 months
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Ask the patient to rate their current level of pain by placing a mark on the line.

SECONDARY OUTCOMES:
Secondary Outcome Measures will be the change of WOMAC Osteoarthritis Index from baseline to posttreatment | 3 months
  Self-administered Western Ontario and McMaster Universities (WOMAC) index is the most common used clinical tools for evaluating patients with knee OA. It includes five questions about pain, two about stiffness, and 17 on degree of disability of activities of daily living.

CONTACTS AND LOCATIONS:
Locations (1):
- Mostafa Bahaa, Damietta, New Damietta, Egypt